CLINICAL TRIAL: NCT06672757
Title: Use of App for Stroke Assessment VS Standard Level of Care During Prehospital Stroke Assessment
Acronym: STRAPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: p-2024-17207
Record Dates: First submitted 2024-08-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Stroke, Acute
Keywords: NIHSS; Paramedic
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Stepped wedge
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention with NIHSS certification and use of app (Experimental): All paramedics who have been NIHSS certified wil be enrolled in this arm. Intervention
  Interventions: Device: CV_AID
- Control - standard operating procedure (No Intervention): Paramedics will remain in this arm until they have been NIHSS certified

INTERVENTIONS:
Device: CV_AID — Upon arrival at the scene, the paramedic utilizes a mobile app with an integrated camera to aid in conducting the National Institutes of Health Stroke Scale (NIHSS) assessment. The app assists in scoring the patient's responses according to NIHSS criteria to determine the severity of stroke symptoms.
  If the app assessment indicates a high likelihood of stroke, transport can be initiated without a conference with the neurovascular centre. The app shares the recorded NIHSS assessment and video of the patient with the neurovascular centre for review.
  While en route, the paramedic confer with the neurovascular centre to discuss the patient's condition and determine appropriate course of action. If the neurovascular centre decides not to treat the patient, transport can be diverted to the nearest hospital.
  The paramedic documents all assessment findings, interventions, and communications related to the stroke patient in the patient care record. U
  Other Names: Education of paramedics
  Arms: Intervention with NIHSS certification and use of app

SUMMARY:
In Denmark, 12,000 people experience a stroke every year. It is the fourth largest cause of death, and costs 4,6 billion Danish crowns in healthcare expenses and lost work income. It is also the leading cause of acquired disability for adults. Pre-hospital recognition of stroke is paramount to ensure fast and correct treatment for patients, in turn leading to better outcomes for patients. As the advanced treatment for ischemic stroke, thrombolysis and thrombectomy, is time-sensitive, even short delays in recognition and treatment can have a large effect on the individual stroke patient.

Paramedics on scene have only a few tools to assist them in recognizing stroke, where clinical scales such as the National Institutes of Health Stroke Scale (NIHSS), Face Arm Speech Time (FAST) or Prehospital Stroke Score (PRESS ) are most commonly used. Despite the use of such instruments, patients with stroke still go unrecognized, and as a result, the unrecognized patient might not be hospitalized, be hospitalized in a hospital without stroke facilities or be hospitalized too late for advanced treatment. Lower quality of communication between paramedics and the stroke centre significantly increases prehospital on-scene time. In a consensus statement from the European Academy of Neurology (EAN) and the European Stroke Organisation (ESO), training paramedics to recognise symptoms of all stroke types was strongly recommended. This study aims to explore whether trained paramedics using a mobile application with NIHSS and video communication to the in-hospital stroke physician may improve triage of acute stroke patients. This intervention will be compared to paramedics using standard procedure and communication through regular channels. It is hypothesized that the number of patients brought to the emergency department with suspected acute stroke and discharged with a stroke diagnosis is significantly higher in the app-group (intervention) compared to standard prehospital model (control).

DETAILED DESCRIPTION:
1. Background 1.1 Stroke In Denmark, 12,000 people experience a stroke every year. It is the fourth largest cause of death, and costs 4,6 billion Danish crowns in healthcare expenses and lost work income. It is also the leading cause of acquired disability for adults.

Pre-hospital recognition of stroke is paramount to ensure fast and correct treatment for patients, in turn leading to better outcomes for patients. As the advanced treatment for ischemic stroke, thrombolysis and thrombectomy, is time-sensitive, even short delays in recognition and treatment can have a large effect on the individual stroke patient. Paramedics on scene have only a few tools to assist them in recognizing stroke, where clinical scales such as the National Institutes of Health Stroke Scale (NIHSS), Face Arm Speech Time (FAST) or Prehospital Stroke Score (PRESS ) are most commonly used. Despite the use of such instruments, patients with stroke still go unrecognized, and as a result, the unrecognized patient might not be hospitalized, be hospitalized in a hospital without stroke facilities or be hospitalized too late for advanced treatment.

A combination of early prehospital identification of stroke, triage to the right level of care and improvement of in-hospital measures to reduce door-to-needle time may result in more patients receiving acute treatment. Lower quality of communication between paramedics and the stroke centre significantly increases prehospital on-scene time. In a consensus statement from the European Academy of Neurology (EAN) and the European Stroke Organisation (ESO), training paramedics to recognise symptoms of all stroke types was strongly recommended.

This study aims to explore whether trained paramedics using a mobile application with NIHSS and digital communication may improve triage of acute stroke patients and ensure the standardised transfer of critical patient data to the in-hospital stroke physician. This intervention will be compared to paramedics using standard procedure with PRESS and communication through regular channels.

Investigators hypothesize that the number of patients brought to the emergency department (ED) with suspected acute stroke and discharged with a stroke diagnosis is significantly higher in the app-group (intervention) compared to standard prehospital model (control).

1.1.1 Incidence and mortality In Denmark, 17.647 patients were registered in 2020 with the diagnosis of Stroke and Transient ischemic attack (TIA) according to the national Danish stroke database DanStroke. Costs of Stroke are expected to increase by 44% by 2040 in Europe. A major part of stroke costs is due to post-stroke need of care due to loss of independency. Acute Stroke revascularization treatment using medical thrombolysis or mechanical endovascular treatment is a critical time-dependent situation as increasing time from symptom onset to start of treatment increases independency for patients post-stroke. Every minute there is a loss of approximately 2 MIO brain cells, hence the term "Time is Brain", and corresponds to more loss of independency in clinical outcome with increasing time from onset of symptoms

1.2 Prehospital assessment of patients with suspected stroke 1.2.1 The potential importance of prehospital assessment A combination of early prehospital identification of stroke, triage to the right level of care and improvement of in-hospital measures to reduce door-to-needle time may result in more patients receiving acute treatment. Lower quality of communication between paramedics and stroke centre significantly increases prehospital on-scene time. As mentioned, the European Academy of Neurology (EAN) and the European Stroke Organisation (ESO) strongly recommend training paramedics to recognise symptoms of all stroke types.

1.3 Current evidence concerning videoassisted prehospital assessment of patients with suspected stroke 1.3.1 Randomized clinical trials PubMed was searched with the search terms "prehospital stroke scales", "prehospital NIHSS", "non-physician NIHSS", "prehospital stroke assessment", "NIHSS in LVO", and "mobile stroke units". The focus was on studies reporting randomised controlled trials, stepped-wedge cluster randomised trials, clinical trials, and cohort studies as well as systematic reviews and meta-analyses of prehospital stroke care. A recent randomised trial, the ParaNASPP trial explored prehospital NIHSS as a common language in the acute stroke chain. This trial showed that introducing prehospital NIHSS with direct communication to the stroke physician, improved care by reducing in-hospital time to CT and by increasing prehospital identification of patients with low NIHSS and subtle symptoms. However, it did not increase diagnostic accuracy.

Another study, the PASTA trial, explored the implementation of a structured protocol and checklists for paramedic stroke assessment to increase thrombolytic rates in a randomised control design. The PASTA checklist was based on structured handover and clinical assessment with a face, arm, speech, time (FAST) test, and concluded that paramedic training in FAST alone did not significantly influence treatment rate. These prehospital stroke scales are usually modified versions of the National Institutes of Health Stroke Scale (NIHSS) and their main purpose is to enable identification of patients with large vessel occlusions (LVOs), eligible for endovascular thrombectomy.

In the PRESTO trial, Duvecot et al. compared the accuracy of eight prehospital stroke scales in detecting LVOs. Since LVOs occur in at most 30% of the general stroke population, most patients have non-LVO stroke with a heterogeneous symptom presentation. The NIHSS is the scale of choice for identification of both LVO and non-LVO strokes. Our literature search did not find any prehospital studies focusing on non-LVO symptoms in minor to moderate strokes. Several in-hospital conducted cohort and inter-rater agreement studies on the NIHSS have shown high levels of agreement when used by non-physicians. No studies considered whether prehospital NIHSS could be implemented in a large-scale prehospital system; however, promising results were presented in cohort studies from the helicopter emergency medical service and mobile stroke units. The prehospital NIHSS studies had poor methodological robustness because of their small sample size and non-randomised design.

1.5 Current practice Currently, paramedics meeting a patient with suspected stroke assess the patients with the PRESS-scale and when deemed necessary the comprehensive stroke centre is contacted, and a teleconference between paramedics and the attending neurologist is initiated. In case of suspected and prehospitally confirmed stroke suspicion, the patient is transported to the comprehensive stroke centre in Roskilde for further evaluation and treatment.

If a stroke is identified at the hospital, it is registered in The Danish Stroke Registry (DanStroke).

ELIGIBILITY:
Inclusion Criteria:

* A. Suspected stroke by paramedic or dispatcher

Exclusion Criteria:

* Technical issues (ie. the telephone does not work, the app does not work).
* Patients who are incarcerated
* Patients seen by a physician prior to assessment by paramedics.
* Subarachnoid Haemorrhage strokes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-10-29 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Prehospital recognition of stroke | From enrollment to patient admission upto 6 hours
  The primary outcome will be prehospital recognition of stroke by paramedics, quantified as the proportion of patients discharged with a final stroke diagnosis who are accepted for stroke evaluation by the neurologist at the neurovascular centre.

SECONDARY OUTCOMES:
Time on scene | From enrollment to the admission upto 6 hours
  Time spent on-scene is a key metric for the evaluation of prehospital health services. Less time spent on scene is directly correlated with time to hospital admittance, presuming correct triage of the patient. As this study introduces a potential delaying factor in the use of an app and the performance of a full NIHSS evaluation, this metric is key to evaluating whether this new initiative is a net positive for patients with stroke.
Door-to-scanner time | From enrollment to the admission upto 12 hours
  Investigators theorise that the availability of a reliable NIHSS score as well as the video material from the evaluation of the patient will enable the neurologist at the neurovascular centre to make faster assessment, which could lead to reduced door-to-scanner times.
Change in 90-day neurological outcome measured by the modified rankin scale (mRS) | 90 days after admission
  The 90-day neurological outcome is important, as this outcome reflects the degree of disability experienced by the patient, and thereby the recovery from stroke. If this study leads to faster and more accurate diagnoses and treatment, investigators to see this reflected in the 90 day-neurological outcome.
  Neurological outcome is measured by the modified rankin scale (mRS), a clinical scale to measure the degree of disability or dependence in daily activities of people who have had a stroke or other neurological diseases. It ranges from 0 (no symptoms) to 6 (death). The mRS is the standard scale for evaluating the patients degree of disability post-stroke, and is available as part of the DanStroke registry data for all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Helle C Christensen, MD, PHD, Principal Investigator — Region Zealand Prehospital Center, Denmark
Locations (1):
- Emergency Medical Services, Næstved, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be completely anonymized according to Danish law before analysis. Due to Danish data regulations, data is not publically available, but access to the registry data used in this project can be applied for by appropriate official channels. Anonymised data from the app can be made available upon reasonable request after the publication of the results.
  All relevant project-related documents will be made available upon reasonable request. Data will be available for any research purpose to all interested parties who have approval from an independent review committee and who have a methodological sound proposal as determined by the steering committee of the current project. Interested parties will be able to request the project specific data by contacting the principal investigator, and registry data by appropriate official channels.

REFERENCES:
- [Background] Gude MF, Blauenfeldt RA, Behrndtz AB, Nielsen CN, Speiser L, Simonsen CZ, Johnsen SP, Kirkegaard H, Andersen G. The Prehospital Stroke Score and telephone conference: A prospective validation. Acta Neurol Scand. 2022 May;145(5):541-550. doi: 10.1111/ane.13580. Epub 2022 Jan 13. PMID 35023151
- [Background] Duvekot MHC, Venema E, Rozeman AD, Moudrous W, Vermeij FH, Biekart M, Lingsma HF, Maasland L, Wijnhoud AD, Mulder LJMM, Alblas KCL, van Eijkelenburg RPJ, Buijck BI, Bakker J, Plaisier AS, Hensen JH, Lycklama A Nijeholt GJ, van Doormaal PJ, van Es ACGM, van der Lugt A, Kerkhoff H, Dippel DWJ, Roozenbeek B; PRESTO investigators. Comparison of eight prehospital stroke scales to detect intracranial large-vessel occlusion in suspected stroke (PRESTO): a prospective observational study. Lancet Neurol. 2021 Mar;20(3):213-221. doi: 10.1016/S1474-4422(20)30439-7. Epub 2021 Jan 7. PMID 33422191
- [Background] Price CI, Shaw L, Islam S, Javanbakht M, Watkins A, McMeekin P, Snooks H, Flynn D, Francis R, Lakey R, Sutcliffe L, McClelland G, Lally J, Exley C, Rodgers H, Russell I, Vale L, Ford GA. Effect of an Enhanced Paramedic Acute Stroke Treatment Assessment on Thrombolysis Delivery During Emergency Stroke Care: A Cluster Randomized Clinical Trial. JAMA Neurol. 2020 Jul 1;77(7):840-848. doi: 10.1001/jamaneurol.2020.0611. PMID 32282015
- [Background] Guterud M, Fagerheim Bugge H, Roislien J, Kramer-Johansen J, Toft M, Ihle-Hansen H, Bache KG, Larsen K, Braarud AC, Sandset EC, Ranhoff Hov M. Prehospital screening of acute stroke with the National Institutes of Health Stroke Scale (ParaNASPP): a stepped-wedge, cluster-randomised controlled trial. Lancet Neurol. 2023 Sep;22(9):800-811. doi: 10.1016/S1474-4422(23)00237-5. PMID 37596006
- [Background] Viereck S, Moller TP, Iversen HK, Christensen H, Lippert F. Medical dispatchers recognise substantial amount of acute stroke during emergency calls. Scand J Trauma Resusc Emerg Med. 2016 Jul 7;24:89. doi: 10.1186/s13049-016-0277-5. PMID 27388490
- [Background] Walter S, Audebert HJ, Katsanos AH, Larsen K, Sacco S, Steiner T, Turc G, Tsivgoulis G. European Stroke Organisation (ESO) guidelines on mobile stroke units for prehospital stroke management. Eur Stroke J. 2022 Mar;7(1):XXVII-LIX. doi: 10.1177/23969873221079413. Epub 2022 Feb 9. PMID 35300251
- [Background] Chiu LQ, Quek DYJ, Salihan RB, Ng WM, Othman RB, Lee CH, Oh DCT. ACT-FAST: a quality improvement project to increase the percentage of acute stroke patients receiving intravenous thrombolysis within 60 minutes of arrival at the emergency department. Singapore Med J. 2021 Sep;62(9):476-481. doi: 10.11622/smedj.2020040. Epub 2020 Mar 31. PMID 32227791
- [Background] Saver JL. Time is brain--quantified. Stroke. 2006 Jan;37(1):263-6. doi: 10.1161/01.STR.0000196957.55928.ab. Epub 2005 Dec 8. PMID 16339467
- [Background] Rudd AG, Bladin C, Carli P, De Silva DA, Field TS, Jauch EC, Kudenchuk P, Kurz MW, Laerdal T, Ong M, Panagos P, Ranta A, Rutan C, Sayre MR, Schonau L, Shin SD, Waters D, Lippert F. Utstein recommendation for emergency stroke care. Int J Stroke. 2020 Jul;15(5):555-564. doi: 10.1177/1747493020915135. Epub 2020 Mar 29. PMID 32223543
- [Background] Wardlaw JM, del Zoppo G, Yamaguchi T. Thrombolysis for acute ischaemic stroke. Cochrane Database Syst Rev. 2000;(2):CD000213. doi: 10.1002/14651858.CD000213. PMID 10796329
- [Background] Berge E, Whiteley W, Audebert H, De Marchis GM, Fonseca AC, Padiglioni C, de la Ossa NP, Strbian D, Tsivgoulis G, Turc G. European Stroke Organisation (ESO) guidelines on intravenous thrombolysis for acute ischaemic stroke. Eur Stroke J. 2021 Mar;6(1):I-LXII. doi: 10.1177/2396987321989865. Epub 2021 Feb 19. PMID 33817340
- [Background] Johnsen SP, Ingeman A, Hundborg HH, Schaarup SZ, Gyllenborg J. The Danish Stroke Registry. Clin Epidemiol. 2016 Oct 25;8:697-702. doi: 10.2147/CLEP.S103662. eCollection 2016. PMID 27843349
- [Background] Kobayashi A, Czlonkowska A, Ford GA, Fonseca AC, Luijckx GJ, Korv J, de la Ossa NP, Price C, Russell D, Tsiskaridze A, Messmer-Wullen M, De Keyser J. European Academy of Neurology and European Stroke Organization consensus statement and practical guidance for pre-hospital management of stroke. Eur J Neurol. 2018 Mar;25(3):425-433. doi: 10.1111/ene.13539. Epub 2018 Jan 12. PMID 29218822
- [Background] Drenck N, Viereck S, Baekgaard JS, Christensen KB, Lippert F, Folke F. Pre-hospital management of acute stroke patients eligible for thrombolysis - an evaluation of ambulance on-scene time. Scand J Trauma Resusc Emerg Med. 2019 Jan 9;27(1):3. doi: 10.1186/s13049-018-0580-4. PMID 30626404
- [Background] Berglund A, Svensson L, Sjostrand C, von Arbin M, von Euler M, Wahlgren N; HASTA Collaborators; Engerstrom L, Hojeberg B, Kall TB, Mjornheim S, Engqvist A. Higher prehospital priority level of stroke improves thrombolysis frequency and time to stroke unit: the Hyper Acute STroke Alarm (HASTA) study. Stroke. 2012 Oct;43(10):2666-70. doi: 10.1161/STROKEAHA.112.652644. Epub 2012 Aug 9. PMID 22879096
- [Background] Mulder MJHL, Jansen IGH, Goldhoorn RB, Venema E, Chalos V, Compagne KCJ, Roozenbeek B, Lingsma HF, Schonewille WJ, van den Wijngaard IR, Boiten J, Albert Vos J, Roos YBWE, van Oostenbrugge RJ, van Zwam WH, Majoie CBLM, van der Lugt A, Dippel DWJ; MR CLEAN Registry Investigators. Time to Endovascular Treatment and Outcome in Acute Ischemic Stroke: MR CLEAN Registry Results. Circulation. 2018 Jul 17;138(3):232-240. doi: 10.1161/CIRCULATIONAHA.117.032600. Epub 2018 Mar 26. PMID 29581124
- [Background] Lees KR, Bluhmki E, von Kummer R, Brott TG, Toni D, Grotta JC, Albers GW, Kaste M, Marler JR, Hamilton SA, Tilley BC, Davis SM, Donnan GA, Hacke W; ECASS, ATLANTIS, NINDS and EPITHET rt-PA Study Group; Allen K, Mau J, Meier D, del Zoppo G, De Silva DA, Butcher KS, Parsons MW, Barber PA, Levi C, Bladin C, Byrnes G. Time to treatment with intravenous alteplase and outcome in stroke: an updated pooled analysis of ECASS, ATLANTIS, NINDS, and EPITHET trials. Lancet. 2010 May 15;375(9727):1695-703. doi: 10.1016/S0140-6736(10)60491-6. PMID 20472172
- [Background] Skajaa N, Adelborg K, Horvath-Puho E, Rothman KJ, Henderson VW, Casper Thygesen L, Sorensen HT. Nationwide Trends in Incidence and Mortality of Stroke Among Younger and Older Adults in Denmark. Neurology. 2021 Mar 30;96(13):e1711-e1723. doi: 10.1212/WNL.0000000000011636. Epub 2021 Feb 10. PMID 33568547
- [Background] Bhatt A. International Council for Harmonisation E6(R2) addendum: Challenges of implementation. Perspect Clin Res. 2017 Oct-Dec;8(4):162-166. doi: 10.4103/picr.PICR_124_17. PMID 29109932